CLINICAL TRIAL: NCT06779552
Title: CardioMEMS HF System Coverage with Evidence Development Study
Status: Recruiting | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: CL1027482
Record Dates: First submitted 2025-01-13; First posted 2025-01-16 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Treatment Group: Heart failure patients implanted with the CardioMEMS PA pressure sensor.
  Interventions: Device: CardioMEMS HF System
- Control Group: Heart failure patients being managed without PA pressure-monitoring.

INTERVENTIONS:
Device: CardioMEMS HF System — PA Pressure Sensor
  Groups: Treatment Group

SUMMARY:
The purpose of the CardioMEMS CED Study is to determine if pulmonary artery (PA) pressure-guided heart failure management using the CardioMEMS™ HF System improves long-term health outcomes in heart failure (HF) patients in the real-world setting.

DETAILED DESCRIPTION:
The CardioMEMS CED Study will assess 2-year HF hospitalization rates and survival for all-cause mortality in heart failure subjects managed with the CardioMEMS HF system, as compared to a contemporaneous control of HF subjects managed without PA pressure-guidance.

ELIGIBILITY:
Inclusion Criteria:

1. Subject implanted with a CardioMEMS pressure sensor (treatment arm only)
2. Subject >=18 years of age at time of implant
3. Subject has a history of acute decompensated HF or HF-related congestion defined by at least one of the following qualifying event types: HF hospitalization, elevated BNP/NT-proBNP

Exclusion Criteria:

1. Subject has history of heart transplant or durable mechanical circulatory device
2. Subject hospitalized with cardiogenic shock or sepsis
3. Subject received prior PA pressure sensor implant (control arm only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include Heart Failure patients in the United States implanted with the CardioMEMS PA pressure sensor and HF patients being managed without PA pressure-monitoring.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-02-07 (Actual); Primary Completion 2032-03 (Estimated); Study Completion 2032-03 (Estimated)

PRIMARY OUTCOMES:
HF Hospitalization Rate. | 2 years
  Compare HF hospitalization rate between the treatment and control groups.

SECONDARY OUTCOMES:
Two-Year Survival | 2 years
  Compare survival between the treatment and control groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Abbott, Pleasanton, California, United States